CLINICAL TRIAL: NCT01990898
Title: Cyclosporine in Interstitial Cystitis: Efficacy, Safety and Mechanism of Action
Acronym: CIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1271
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2016-10

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclosporine (Experimental): Drug: Cyclosporine, Pill form, dosage calculated upon patient study visit, frequency - twice daily, duration - 3 months.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — Drug will be provided to patient's at study visit. Drug is to be taken twice daily. Dosage will be calculated at study visit and provided to patient.
  Other Names: Gengraf Cyclosporine

SUMMARY:
This is a study for patients that have a condition called Interstitial Cystitis, also known as Painful Bladder Syndrome. Patients would have tried at least two different therapies, unsuccessfully,(eg. medications, pelvic floor physical therapy)

The purpose of this research project is to study the immunosuppressive drug Cyclosporine in patients with Interstitial Cystitis to assess how well it works, what the side effects are and what is its mechanism of action. Cyclosporine is a drug that is FDA-approved to prevent organ rejection after kidney, liver, and heart transplant but is not approved by the FDA for Interstitial Cystitis. Several research studies have been published showing that Cyclosporine can improve the symptoms of Interstitial Cystitis, that it works better than a placebo ("sugar pill" or inert treatment) and that it works more effectively than Pentosan Polysulfate (Elmiron), which is an FDA approved therapy. The dose of Cyclosporine used in these studies on Interstitial Cystitis are much lower that the doses used to prevent rejection in transplant patients.

Based on these studies, the American Urological Association has recently published treatment guidelines that recommend Cyclosporine therapy for Interstitial Cystitis after the failure of other more conservative therapies and medications. Nevertheless, much is not known about using Cyclosporine therapy for Interstitial Cystitis including the mechanism of action, the ideal dose, how best to monitor for side effects and in particular whether kidney damage can occur at the low doses used in these studies. In this study, to examine the mechanism of action, blood and urine samples will be collected before, during and after therapy to look at "biomarkers", chemical substances that can be associated with inflammation and tissue injury. We will also test effects of therapy on skin sensation and pain perception because the molecule which Cyclosporine binds to (calcineurin) is also found in nerves that conduct pain signals.

This study is only being done at the Cleveland Clinic and will involve about 30 patients with Interstitial Cystitis.

DETAILED DESCRIPTION:
Based on these studies, the American Urological Association has recently published treatment guidelines that recommend Cyclosporine therapy for Interstitial Cystitis after the failure of other more conservative therapies and medications. Nevertheless, much is not known about using Cyclosporine therapy for Interstitial Cystitis including the mechanism of action, the ideal dose, how best to monitor for side effects and in particular whether kidney damage can occur at the low doses used in these studies. In this study, to examine the mechanism of action, blood and urine samples will be collected before, during and after therapy to look at "biomarkers", chemical substances that can be associated with inflammation and tissue injury. We will also test effects of therapy on skin sensation and pain perception because the molecule which Cyclosporine binds to (calcineurin) is also found in nerves that conduct pain signals.

This study is only being done at the Cleveland Clinic and will involve about 30 patients with Interstitial Cystitis.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18
2. able to give consent
3. commitment to return for follow up appointments
4. agree to all parts of the study, including pain sensation testing
5. total Interstitial Cystitis Symptom Index (ICSI) score >9

Exclusion Criteria:

1. active cancer
2. history of pelvic radiation
3. history of previous urological malignancy
4. serum Cr > 1.5 mg/dl
5. diagnosis of diabetes mellitus types I or II
6. untreated hypertension or blood pressure on treatment > 140/90
7. proteinuria at enrollment
8. current or previous urinary diversion or bladder augmentation
9. chronic use of a medication class with significant impact on Cyclosporine A (CyA) blood levels (eg. macrolide antibiotics, phenytoin, oral antifungals, calcium channel blockers)
10. untreated urinary tract infection
11. pregnant or breast feeding
12. neurological impairment or spinal cord injury
13. known hypersensitivity to CyA
14. concurrent use of another immunosuppressive drug (eg. oral corticosteroids, tacrolimus, mycophenolate mofetil)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Shoskes, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic - Main Campus Only, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Cyclosporine
Period: Overall Study
Arm/Group | Treatment
Started | 26
3 Months | 22
Completed | 22
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 50 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Symptom Improvement of Interstitial Cystitis
Description: Number of participants with > 30% Improved Interstitial Cystitis Symptoms Index (ICSI) which is measured on a scale from 0 - 19 where the higher numbers are worse. No additional analyses have been done.
Time Frame: 3 Months
Measure: Number; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 22
Participants | 9

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 2/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=26)
Hypertension (Cardiac disorders) | 1
Elevated Serum Glucose (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No